CLINICAL TRIAL: NCT07217860
Title: A Multicenter, Long-term, Open-Label, Safety, Tolerability, and Efficacy Study of Azetukalner in Bipolar I or II Depression
Brief Title: An Open-label Study of Azetukalner in Bipolar I or II Depression (X-CEED-OLE)
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XPF-010-B302
Record Dates: First submitted 2025-10-14; First posted 2025-10-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Depression; Bipolar I Disorder; Bipolar Disorder; Bipolar II Disorder
Keywords: Bipolar; XEN1101; Azetukalner
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azetukalner 20 mg (Experimental)
  Interventions: Drug: Azetukalner

INTERVENTIONS:
Drug: Azetukalner — Azetukalner 20 mg taken orally once a day with food (with the evening meal when possible) for 52 weeks.

SUMMARY:
X-CEED-OLE is a Phase 3, multicenter, open-label study to evaluate the long-term safety, tolerability, and efficacy of azetukalner in adult participants who successfully completed an antecendent Phase 3 azetukalner bipolar depression study.

ELIGIBILITY:
Inclusion Criteria:

* Participant successfully completed the treatment period in a Phase 3 antecedent study evaluating azetukalner in participants with bipolar depression.
* Participant provides written informed consent to participate in the study, is able to understand the procedures and study requirements, and agrees to abide by them.
* Participant is willing to comply with the contraception requirements.

Exclusion Criteria:

* Participant met any of the withdrawal criteria, discontinued study drug early, or was terminated early from an antecedent study.
* Participant had any protocol deviations in an antecedent study that, in the opinion of the investigator, would preclude participation in this study.
* Participant has any medical condition, personal circumstance, or ongoing AE (from an antecedent study) that, in the opinion of the investigator, exposes the participant to unacceptable risk by participating in the study or prevents adherence to the protocol.
* Participant is pregnant, breastfeeding, or planning to become pregnant.
* Participant is planning to enter a clinical study with a different investigational drug or planning to use any experimental device for the treatment of any medical condition during the study or within 28 days after completion of this study.
* Participant is judged by the investigator to have a significant risk for self-harm or suicidal behavior during their participation in the study or is considered to be an imminent danger to themself or others.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Severity and frequency of treatment-emergent adverse events, serious adverse events, adverse events of special interest, and events of clinical interest | From the start of treatment in the open-label extension study through 8 weeks after the last dose

SECONDARY OUTCOMES:
Change from baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score over time | From baseline through the active extension treatment (Week 52)
Change in Clinical Global Impression of Severity (CGI-S) score over time | From baseline through the active extension treatment (Week 52)
Change from baseline in the Snaith-Hamilton Pleasure Scale (SHAPS) total score over time | From baseline through the active extension treatment (Week 52)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - CenExel iResearch, Decatur, Georgia
  - Lumina Clinical Research Center, Cherry Hill, New Jersey
  - Clinical Neuroscience Solutions Memphis, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Randomized Study of Azetukalner Versus Placebo in Depressive Episodes Associated With Bipolar I or II Disorder (Bipolar Depression) (X-CEED) — https://www.clinicaltrials.gov/study/NCT07172516?intr=XEN1101&page=2&rank=13